CLINICAL TRIAL: NCT02677389
Title: Active Living After Cancer: Building a Physical Activity Intervention Into Clinical Care for Breast and Colorectal Cancer Survivors in Wisconsin
Brief Title: Survivorship Care Plan in Promoting Physical Activity in Breast or Colorectal Cancer Survivors in Wisconsin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW15059; NCI-2016-00111 (Registry Identifier: NCI Trial ID); 2015-1295 (Other: Institutional Review Board); A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison)
Record Dates: First submitted 2016-02-01; First posted 2016-02-09 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-02

CONDITIONS: Cancer Survivor; Healthy Subject; Stage I Colorectal Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIA Colorectal Cancer; Stage IIB Breast Cancer; Stage IIB Colorectal Cancer; Stage IIC Colorectal Cancer; Stage IIIA Breast Cancer; Stage IIIA Colorectal Cancer; Stage IIIB Breast Cancer; Stage IIIB Colorectal Cancer; Stage IIIC Breast Cancer; Stage IIIC Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Enhanced SCP) (Experimental): See Detailed Description
  Interventions: Other: Educational Intervention; Other: Internet-Based Intervention; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (SCP) (Active Comparator): Participants receive a standard SCP, comprised of a treatment and follow up recommendations, including basic physical activity guidance, copy of the USDA Dietary Guidelines for Americans, as well as standardized emails with wellness tips and information on stress management provided from the American Heart Association's website on "Healthy Habits" at 1, 2, 4, and 8 weeks. Specific topics in emails include "positive self-talk", "daily relaxation breathing techniques", "better sleep", and "ways to find pleasure".
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational material regarding physical activity and standardized emails with wellness tips and information on stress management
  Other Names: Education for Intervention; Intervention, Educational
Other: Internet-Based Intervention — Receive email and technical or how-to support from study coordinator
  Arms: Arm I (Enhanced SCP)
Device: Monitoring Device — Wear a Fitbit web-integrated physical activity tracker
  Other Names: Monitor; Fitbit
  Arms: Arm I (Enhanced SCP)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies how well survivorship care plan works in promoting technology-based physical activity in breast or colorectal cancer survivors in Wisconsin. A survivorship care plan may help doctors to better understand how they can help people who have been diagnosed with cancer to become more physically active. It is not yet known whether a standardized cancer survivor plan used as part of routine care or a technology-based physical activity intervention is better in promoting physical activity in breast or colorectal cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the feasibility of enrolling breast and colorectal cancer survivors along with a co-survivor into a randomized physical activity promotion trial.

II. Determine the short-term effect of an enhanced survivorship care plan (SCP) compared to the standard SCP on objectively-measured physical activity among survivors and co-survivors.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (Enhanced SCP): Participants receive an enhanced SCP, comprised of a personalized document that summarizes treatment and follow up recommendations, including basic physical activity guidance. Participants also receive a copy of the United States Department of Agriculture (USDA) Dietary Guidelines for Americans, as well as standardized emails with wellness tips and information on stress management provided from the American Heart Association's website on "Healthy Habits" at 1, 2, 4, and 8 weeks. Specific topics in emails include "positive self-talk", "daily relaxation breathing techniques", "better sleep", and "ways to find pleasure". Participants also wear a Fitbit web-integrated physical activity tracker daily for 12 weeks and receive email feedback specific to each participant based on a series of factors, including their Fitbit data, Emails may provide encouragement, such as "keep up the good work", and/or very specific instructions regarding compliance with the intervention, goals for meeting physical activity goals, potential strategies to increase/maintain levels of physical activity, etc., and technical or how-to support including how to use the device and website, or questions about goal-setting.

ARM II (Control): Participants receive a standard SCP, comprised of a personalized document that summarizes treatment and follow up recommendations, including basic physical activity guidance. Participants also receive a copy of the USDA Dietary Guidelines for Americans, as well as standardized emails with wellness tips and information on stress management provided from the American Heart Association's website on "Healthy Habits" at 1, 2, 4, and 8 weeks. Specific topics in emails include "positive self-talk", "daily relaxation breathing techniques", "better sleep", and "ways to find pleasure".

ELIGIBILITY:
Inclusion Criteria:

* CRITERIA FOR SURVIVORS:

  * Have a diagnosis of stage I-III female breast cancer or colorectal cancer within the past 5 years; bilateral or multiple primary breast cancers are permitted; individuals who have had more than one type of cancer (e.g., both breast and melanoma) are permitted as long as the breast (or colorectal) diagnosis meets the other criteria and primary treatment for any cancer is not ongoing
  * Have completed primary treatment for their cancer; primary treatment will be defined as having completed all (a) definitive cancer surgery, (b) (neo)adjuvant chemotherapy, and/or (c) (neo)adjuvant radiation; breast cancer patients still receiving adjuvant endocrine or human epidermal growth factor receptor 2 (HER2) targeted therapies are eligible, as would colon cancer patients receiving a targeted agent; if there is any question whether a patient meets this eligibility requirement, Dr. Tevaarwerk (co-I, Oncology) will adjudicate
  * Are willing to attempt increase in physical activity level
  * Have a co-survivor (friend or family member) willing to participate in this research study
* ELIGIBILITY CRITERIA FOR BOTH SURVIVORS AND CO-SURVIVORS:

  * Have high-speed access to the internet at home or work; This could be broadband, digital subscriber line (DSL), and/or access on a smartphone or tablet via a wireless provider
  * Fluent in English
  * Willing and able to attend study visits at the University of Wisconsin (UW) - Madison
  * Co-survivors must be over the age of 18 years

Exclusion Criteria:

* EXCLUSION CRITERIA SPECIFIC TO SURVIVORS:

  * Survivors must not have evidence of recurrent or metastatic disease
  * Survivors must not have previously received an SCP or are unwilling to receive one
  * Survivors must not be performing >= 100 minute (min)/week of moderate-vigorous physical activity
* EXCLUSION CRITERIA FOR BOTH SURVIVORS AND CO-SURVIVORS:

  * Conditions that would interfere with the safety of moderate-to-vigorous intensity physical activity; participants will be screened for safety using the validated Physical Activity Readiness Questionnaire (PAR-Q)
  * Any physical or mental health condition that would interfere with full participation in the study, including individuals who are unable to read consent materials or appear to lack the capacity to consent
  * Any individual considered to be that of a "vulnerable group", including pregnant women and prisoners

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Feasibility as defined by recruitment rate | Up to 12 weeks
  Measures include recruitment rate (ability to recruit ≥5 patients per month to the study), retention rate (ability to collect all measures on ≥80% of randomized patients) and patient satisfaction with SCP, Fitbit, and physical activity intervention materials, both overall and by cancer type (breast/colon).

SECONDARY OUTCOMES:
Physical activity as measured by the ActiGraph GT3X+ accelerometer (Arm I) | Up to 12 weeks
  ActiGraph accelerometer will be compared between the arms (intervention and control) using a mixed effects model for repeated daily measures at week 0 (baseline) and week 12. Explanatory factors will be study week, measurement day and the randomization group by week interaction (the primary parameter of interest).
Physical activity as measured by the ActiGraph GT3X+ accelerometer (Arm II) | Up to 12 weeks
  ActiGraph GT3X+ accelerometer will be compared between the arms (intervention and control) using a mixed effects model for repeated daily measures at week 0 (baseline) and week 12. Explanatory factors will be study week, measurement day and the randomization group by week interaction (the primary parameter of interest).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cadmus-Bertram, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Rastogi S, Tevaarwerk AJ, Sesto M, Van Remortel B, Date P, Gangnon R, Thraen-Borowski K, Cadmus-Bertram L. Effect of a technology-supported physical activity intervention on health-related quality of life, sleep, and processes of behavior change in cancer survivors: A randomized controlled trial. Psychooncology. 2020 Nov;29(11):1917-1926. doi: 10.1002/pon.5524. Epub 2020 Oct 4. PMID 32808383
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/